CLINICAL TRIAL: NCT02782702
Title: Evaluation of the Improvement of Quality of Life of Patients Suffering From Hailey Hailey or Darier Disease After Injections of Botulism Toxin Into Large Folds. Toxin Hailey Darier
Brief Title: Evaluation of the Improvement of Quality of Life of Patients Suffering From Hailey Hailey or Darier Disease After Injections of Botulism Toxin Into Large Folds.
Acronym: ToxHD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14 7316 02
Record Dates: First submitted 2016-05-20; First posted 2016-05-25 (Estimated); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Hailey-Hailey Disease; Darier Disease
Keywords: Botulism Toxin
MeSH Terms: conditions — Pemphigus, Benign Familial; Darier Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Botulism Toxin treatment (Experimental): Injection of 50 UI Botulism toxin for the treated zone
  Interventions: Drug: Botulism Toxin Treatment

INTERVENTIONS:
Drug: Botulism Toxin Treatment — Injection of 50 UI of botulism toxin for treated zone

SUMMARY:
Hailey Hailey and Darier disease are rare genetic dermatoses. Mutations of 2 genes (ATP2C1 or ATP2A2 respectively) are responsible for the diseases. These genes have a key role in calcium pump; their defect create abnormal link between keratinocytes' desmosomes and induce skin lesions. Clinically, patients present with inflammatory lesions located in the folds. Quality of life is impaired because of pain, pruritus and tendency to infections. Lesions are permanent but acute exacerbations occur in hot seasons because of increased sweating. Usual therapies are often not effective (local treatment, laser, phototherapy). Because sweating is a well established inducing or aggravating factor, botulism toxin could be an effective treatment for these diseases.

Botulism toxin is already used in clinical practice and acts via a decreased sweet secretion. Improvement of skin lesions in Hailey-Hailey or Darier diseases has been previously reported in a few cases but there is no study properly evaluating the benefit of such treatment.

The aim of the project is to study the improvement of quality of life for patients suffering from Hailey-Hailey or Darier diseases after a injections of botulism toxin in large skin folds. The principal objective is to estimate the distribution of the variation of quality of life at M1 vs. baseline.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis (clinical and histological features) of Hailey Hailey or Darier diseases.
* Moderate to very severe lesions located in large folds
* Patient aged 18 ans or more
* Patient with health coverage
* Patient who have signed the consent form
* Patient proficient into filling out the questionnaires.

Exclusion Criteria:

* Hypersensibility to toxin or excipients
* Myastheny
* Deglutition's problems
* Past medical history of dysphagia or aspiration pneumonia
* Pregnancy (positive B-HCG test performed a maxima 72h before) or breastfeeding
* Mental , physical incapacity to fill in the questionnaires
* Guardianship patients
* Skin infections at the inclusion visit
* Application in the last 7 days at the site of injection of local treatments (apart emollients or antiseptics) or injections of botulism toxin or dynamic phototherapy or laser in the last 6 months.
* Systemic treatment with aminosides in the last 15 days
* Inclusion in another study in the last 2 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of quality of life measured by change in the DLQI score | Day 0 and day 30
  Variation of DLQI score between Baseline and M1

SECONDARY OUTCOMES:
Evaluation of quality of life measured by change in the DLQI score | Day 0 and day 90
  Variation of DLQI score between Baseline and M3
Evaluation of quality of life measured by change in the DLQI score | Day 0 and day 180
  Variation of DLQI score between Baseline and M6
Evaluation of skin improvement in treated areas using change the IGA score | Day 0 and Day 30
  Variation of IGA score between Baseline and M1
Evaluation of skin improvement in treated areas using change the IGA score | Day 0 and Day 90
  Variation of IGA score between Baseline and M3
Evaluation of skin improvement in treated areas using change the IGA score | Day 0 and Day 180
  Variation of IGA score between Baseline and M6
Evaluation of psychosocial impairment at measured by change in the HidroQoL score | Day 0 and Day 30
  Variation of HidroQoL score between Baseline and M1
Evaluation of psychosocial impairment measured by change in the HidroQoL score | Day 0 and Day 90
  Variation of HidroQoL score between Baseline and M3
Evaluation of psychosocial impairment measured by change in the HidroQoL score | Day 0 and Day 180
  Variation of HidroQoL score between Baseline and M6
Evaluation by the investigator of the treated lesions global severity change as assessed by comparison using measurement of the affected area | Day 0 and Day 30
  Variation of treated lesions severity between Baseline and M1
Evaluation by the investigator of the treated lesions global severity change as assessed by comparison using measurement of the affected area | Day 0 and Day 90
  Variation of treated lesions severity between Baseline and M3
Evaluation by the investigator of the treated lesions global severity change as assessed by comparison using measurement of the affected area | Day 0 and Day 180
  Variation of treated lesions severity between Baseline and M6
Evaluation of patient's satisfaction Using the IGA score " Improvement Global Assessment " | Day 180
Evaluation of patient treatment acceptability using visual analogic pain scale | Day 0 after injection
Evaluation of acceptability over the medium to long term as assessed by occurence of side effects | Day 30
Evaluation of acceptability over the medium to long term as assessed by occurence of side effects | Day 90
Evaluation of acceptability over the medium to long term as assessed by occurence of side effects | Day 180
Evaluation of long term efficacy as assessed by percentage of non-responder patients with IGA score egal to 0 | Day 30
Evaluation of long term efficacy as assessed by delay for significant relapse (reappearance of skin lesions justifying treatment) | Up to 180 days
Evaluation of long term efficacy as assessed by comparison between the number of infection episodes occurred during the 6 months before the study or during the 6 months of the study | Up to 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Aude MAZA RIOLAND, MD, Principal Investigator — University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dreyfus I, Maza A, Rodriguez L, Merlos M, Texier H, Rousseau V, Sommet A, Mazereeuw-Hautier J. Botulinum toxin injections as an effective treatment for patients with intertriginous Hailey-Hailey or Darier disease: an open-label 6-month pilot interventional study. Orphanet J Rare Dis. 2021 Feb 18;16(1):93. doi: 10.1186/s13023-021-01710-x. PMID 33602313